CLINICAL TRIAL: NCT01775241
Title: Sleep Apnoea Syndrome Without Chronic Heart Failure
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 10-080
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Sleep Apnoea Syndrome
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
It is the objective of this study to collect scientific data of sleep apnoea syndrome patients´ cardiac and respiratory function by additional sensors.

ELIGIBILITY:
Inclusion Criteria:

* patients with supected sleep apnoea syndrome and scheduled diagnosis at a sleep laboratory
* male and female patients aged at least 18 years
* persons who understand and follow the instructions of the study staff
* singed informed consent

Exclusion Criteria:

* persons being housed in an institution by court or governmental order
* pregnancy or breastfeeding
* patients who are not able to consent
* acute or chronic inflammations of the external and middle auditory canal
* abnormal anatomic proportionsof the external and middle auditory canal which are pathological or congenital, for example limitation of the auditory canal
* persons in a dependence or in an employment contract to the investigator
* participation in another study at the same time

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with or with supected sleep apnoea syndrome
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2011-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Data collection | 1 night

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy Hospital Aachen, Aachen, North Rhine Westfalia, Germany